CLINICAL TRIAL: NCT01194960
Title: A Randomized Phase II Study to Assess the Activity of TroVax® (MVA-5T4) Plus Docetaxel Versus Docetaxel Alone in Subjects With Progressive Hormone Refractory Prostate Cancer
Brief Title: TroVax® In Subjects With Hormone Refractory Prostate Cancer (HRPC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Collaborators: MedSource LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV2/001/09
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: cancer of prostate; cancer of the prostate; neoplasms prostate; neoplasms prostatic; prostate cancer; prostate neoplasms; prostatic cancer; prostate specific antigen; prostatic hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Docetaxel; TroVax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel Alone (Active Comparator): Subjects will receive 10 cycles of Docetaxel alone until toxicity or progression.
  Interventions: Drug: Docetaxel
- TroVax plus Docetaxel (Experimental): Subjects will receive both TroVax plus 10 cycles of Docetaxel.
  Interventions: Drug: Docetaxel; Drug: TroVax

INTERVENTIONS:
Drug: Docetaxel — Subjects will receive 10 cycles of Docetaxel alone until toxicity or progression.
Drug: TroVax — Trovax on Days 1,10, 22 and then Weeks 7, 10, 13, 19, 25, 31 and 37
  Arms: TroVax plus Docetaxel

SUMMARY:
Based on both pre-clinical and clinical data, it may be advantageous to administer a cancer vaccine before chemotherapy to enhance immune responses, thus leading to a more effective therapeutic approach for subjects with metastatic HRPC. This clinical study will evaluate the role of combination therapy of TroVax® plus Docetaxel vs. Docetaxel alone on the progression free survival (PFS) of subjects with HRPC.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Signed & dated written informed consent obtained from subject in accordance w/local regulations.
2. Histologically confirmed conventional and/or mucinous adenocarcinoma of the prostate. If histological confirmation is not available, cytological confirmation will be permitted in lieu.
3. Must meet one of following 3 criteria for progressive disease following androgen deprivation:

A. Subjects w/nodal or visceral metastases:

Must have progressive disease defined by RECIST criteria or defined by the Prostate Cancer Clinical Trials Working Group II (Scher et al. 2008).

B. Subjects w/no measurable disease:

PSA only disease must have an elevated PSA as defined by Consensus Criteria Prostate Cancer Clinical Trials Working Group II (Scher et al. 2008). PSA must indicate progressive disease defined as rising PSA values, at least 7 days apart, >2 ng/mL in the 28 days prior to randomization.

C. Subjects w/bone involvement:

New disease on bone scan as defined by Consensus Criteria Prostate Cancer Clinical Trials Working Group II (Scher et al. 2008). 4. Subjects on stable dose of bisphosphonates showing subsequent tumor progression may continue on this medication; however, subjects are not allowed to initiate bisphosphonate therapy w/in 28 days prior to starting study treatment at Week 1 or at any time after that during the study, 5. Must be clinically immunocompetent. Clinical immunocompetence assumed unless subject has been diagnosed as immunosuppressed, is receiving immunosuppressive chemotherapy for oncology disorders, or is receiving immunosuppressive therapy following transplant, in which case they will be excluded.

6. Subject free of clinically apparent/active autoimmune disease (no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's Disease, Hashimoto's Thyroiditis, Multiple Sclerosis, & Rheumatoid Arthritis).

7. Subject has adequate bone marrow function defined by Absolute Lymphocyte Count (ALC) ≥ 500/µL, Absolute Neutrophil Count (ANC) >1200/µL, Platelet Count >100,000/µL.

8. Subject has peripheral neuropathy grade ≤1. 9. Subject has ECOG status of 0 or 1. 10. Minimum life expectancy ≥6 months. 11. Progressive disease (as defined above) must be documented after discontinuation of the hormonal and anti-androgen therapy.

12. Subject continues to stay on medical treatment such as LHRH agonists or LHRH antagonists to maintain testosterone value of <50ng/dL.

EXCLUSION CRITERIA:

1. Subject has received prior chemotherapy for prostate cancer at any time. Subject has received chemotherapy for any other reason within five years of screening.
2. Subject is receiving any other hormonal therapy, including any dose of Megestrol Acetate, Finasteride, any herbal product known to decrease PSA levels (e.g., Saw Palmetto & PC-SPES), or any systemic corticosteroid must discontinue agent for at least 4 weeks prior to the anticipated Week 1 visit. LHRH agonists or LHRH antagonists do not need to be discontinued.
3. Subject has started bisphosphonate or denosumab therapy less than 28 days before the anticipated Week 1 visit.
4. Subject is using supplements or complementary medicines/botanicals. Subjects should review label w/their doctor prior to enrolment. Exceptions to this exclusion:

   * Conventional multivitamin supplements
   * Selenium
   * Lycopene
   * Soy supplements
   * Vitamin E
   * Fish oil supplements
   * Vitamin D
   * Glucosamine supplements
   * Age-related eye disease vitamins
   * Ginkgo biloba
5. Subject has had major surgery or radiation therapy completed <4 weeks prior to screening.
6. Corticosteroids are not permitted except for (a) nasal sprays and inhalers, (b) orally prescribed as replacement therapy in the case of adrenal insufficiency, (c) oral or IV dexamethasone administration used acutely in combination with docetaxel, (d) parenteral use on a single occasion, (e) low dose parenteral use for a maximum of 5 days and (f) acute and sporadic parenteral use for acute asthma.
7. Subject is known to test positive for HIV or hepatitis B or C.
8. Subject receiving concurrent chemotherapy, immunotherapy, radiotherapy or investigational agents.
9. Subject has Platelet count >400,000/μL; Monocytes >80,000/μL; Haemoglobin <11g/dL.
10. Subject has cerebral metastases (known from previous investigations or clinically detectable).
11. Subject has serum testosterone >50ng/dL.
12. Subject has rheumatoid disease (asymptomatic subjects w/controlled & rarely flaring rheumatoid arthritis are also excluded).
13. Subject exhibits evidence of symptomatic congestive heart failure, pulmonary embolus, vascular thrombosis, transient ischemic attack, cerebrovascular accident, unstable angina, myocardial infarction or active ischemia on ECG. If an ECG taken prior to screening but within 28 days of the anticipated Week 1 visit is not available, an ECG must be performed at screening.
14. Subject has uncontrolled severe hypertension >150/100mm Hg (if controlled w/medication this is not an exclusion).
15. Subject is hypotensive.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Week 37
  To establish whether the incidence of progression-free survival (as defined by the absence of progression assessed by both RECIST and PCWG2 criteria) at week 37 in the TroVax® plus Docetaxel treatment arm is higher than the incidence in the Docetaxel alone treatment arm.

SECONDARY OUTCOMES:
Clinical progression-free survival | 37 weeks
  To establish whether the incidence of clinical progression-free survival (defined by the absence of progression assessed by RECIST criteria alone) at week 37 in the TroVax® plus Docetaxel treatment arm is higher than the incidence in the Docetaxel alone treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anna C. Ferrari, MD, Principal Investigator — New York University Cancer Institute
Locations (7):
- United States (7):
  - San Bernardino Urology, San Bernardino, California
  - Stanford University Medical Center, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - GU Research Network, Omaha, Nebraska
  - New York University Cancer Institute, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Charleston Hematology Oncology Associates, Charleston, South Carolina

REFERENCES:
- [Result] Harrop R, Chu F, Gabrail N, Srinivas S, Blount D, Ferrari A. Vaccination of castration-resistant prostate cancer patients with TroVax (MVA-5T4) in combination with docetaxel: a randomized phase II trial. Cancer Immunol Immunother. 2013 Sep;62(9):1511-20. doi: 10.1007/s00262-013-1457-z. Epub 2013 Jul 23. PMID 23877659